CLINICAL TRIAL: NCT04327882
Title: Interest of Clinical Ultrasound in Patients Consulting for Dyspnea in the Emergency Department: an Observational Bicentric Study
Brief Title: Point-of-care Ultrasound Interest in Dyspneic Emergency Department Patients: an Observational Bicentric Study
Acronym: ECUDYS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Principal Investigator, Xavier Bobbia, Doctor, Centre Hospitalier Universitaire de Nīmes
Other Study IDs: XBobbia/ECUDYS
Record Dates: First submitted 2020-03-27; First posted 2020-03-31 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Dyspnea
Keywords: Point-of-care system; Ultrasonography; Dyspnea
MeSH Terms: conditions — Dyspnea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Point-of-care ultrasound — performance of a POCUS: lung and cardiac ultrasound mainly

SUMMARY:
The diagnostic value of Point-of-care ultrasound (POCUS) in emergency department (ED) dyspneic patients is shown by numerous studies with a limited number of patients. Recently, Zanobetti et al. showed the POCUS diagnostic performance in dyspneic patients in 2600 patients. This study was monocentric and few physicians performed the ultrasounds. Moreover they were experts. The POCUS diagnostic performance performed in a large number of dyspneic ED patients by many physicians with heterogeneous experience is not known. The investigators are carrying out a bicentric study in two large medical teams routinely practicing POCUS. The main objective of this study is to show the diagnostic concordance between the diagnosis resulting from the POCUS results in emergency department dyspneic patients and the diagnosis of discharge from the emergency department in a large medical team with a heterogeneous level of training and experience. The secondary objective is to study these different diagnostic concordances according to the level of ultrasound expertise of the ER practitioners.

DETAILED DESCRIPTION:
* Status of the issue and objective of the research Emergency Clinical Ultrasound (ECU) has shown excellent diagnostic relevance in patients presenting to emergency departments for dyspnea. A recent study including more than 2600 dyspneic patients in the emergency department shows that the diagnosis made with the ECU alone has a good concordance with the diagnosis of end of management in the emergency department but with a significantly shorter duration of obtaining it (186 ± 72 min vs 24 ± 10 min p = 0.025). This study, like many on the ECU, shows good performance when ultrasound is performed by experts. Confirmation that the ECU has a diagnostic performance comparable to all the examinations performed in the standard management of dyspneic patients, when applied by a large team of emergency physicians, is a necessity. The main objective of this study is to show the diagnostic concordance between the diagnosis resulting from the results of the ECU in dyspneic patients in the emergency department and the diagnosis at discharge from the emergency department in a large medical team with a heterogeneous level of training and experience. The secondary objective is to study these different diagnostic concordances according to the level of ultrasound expertise of the ER practitioners.
* Population :

Adult patients (> 18 years old) admitted to the emergency department for a main reason of dyspnea.

- Method of observation : This will be a prospective bicentric observational study.

* Origin and nature of nominative data collected. Data collected from computerized patient records.
* Mode of data flow The data collected will be noted on an anonymized Excel file for analysis.
* Duration and organization of the research Expected duration: 2 years, including an 18-month inclusion period to allow for the inclusion of 2600 patients. Data is collected by the trial investigators.
* Method of data analysis Descriptive statistical analysis and comparison of concordance between different diagnostic methods
* Justification of the number of subjects or power analysis. 2600 to allow comparison with the original publication.

ELIGIBILITY:
Inclusion Criteria:

* Primary reason for emergency Department admission is dyspnea

Exclusion Criteria:

* Pregnant or breastfeeding women
* Persons not benefiting from a social security scheme
* Persons deprived of liberty
* Patient participates in another study
* The patient is in a period of exclusion determined by a previous study.
* The patient is under legal protection, guardianship or trusteeship.
* Patient refuses to participate
* It proves impossible to give informed information about the subject matter
* The patient is not fluent in French.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients managed in both investigative emergency departments whose primary reason for management is dyspnea may be included. Patients with POCUS are included.
Sampling Method: Non-Probability Sample
Enrollment: 2600 (Estimated)
Dates: Start 2019-09-16 (Actual); Primary Completion 2021-03-16 (Estimated); Study Completion 2021-09-16 (Estimated)

PRIMARY OUTCOMES:
Diagnostic concordance | Day 1
  Diagnostic concordance between the POCUS diagnosis in emergency department dyspneic patients and the emergency department discharge diagnosis

SECONDARY OUTCOMES:
Diagnostic concordance and expertise | Day 1
  Diagnostic concordances based on the level of ultrasound expertise of emergency department practitioners
Diagnostic performance of each ultrasound tool | Day 1
  Diagnostic performance of each ultrasound tool used: each pulmonary ultrasound profile, each echocardiographic evaluation or measurement.
Prognostic performance of each ultrasound tool | Day 1
  Prognostic performance of each ultrasound tool used: each pulmonary ultrasound profile, each echocardiographic evaluation or measurement.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hôpital La Timone, Marseille
  - CHU Nîmes, Nîmes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vauthier C, Chabannon M, Markarian T, Taillandy Y, Guillemet K, Krebs H, Bazalgette F, Muller L, Claret PG, Bobbia X. Point-of-care chest ultrasound to diagnose acute heart failure in emergency department patients with acute dyspnea: diagnostic performance of an ultrasound-based algorithm. Emergencias. 2021 Dec;33(6):441-446. English, Spanish. PMID 34813191